CLINICAL TRIAL: NCT05867758
Title: Addressing Social Isolation, Loneliness and Promoting Psychological Wellbeing in International Students
Brief Title: Psychosocial Blended Group Intervention RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-11-22
Record Dates: First submitted 2022-11-21; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2022-11

CONDITIONS: Social Isolation
Keywords: social isolation; international college students; loneliness; psychosocial group intervention; blended intervention
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial of a Group intervention with international college students
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Group of participants (9 to 12) participating in the psychosocial group intervention (8 sessions, one per week) and receiving the self-help digital materials each week.
  Interventions: Other: Psychosocial group intervention
- Control group - waiting list (No Intervention): Group of participants (9 to 12) receiving the self-help digital materials each week, who will take part in the psychosocial group intervention once the data collection will be over

INTERVENTIONS:
Other: Psychosocial group intervention — The psychosocial group intervention is composed of 8 weekly sessions of 90 minutes each and the receiving of self-help digital materials. Both organized as following: 2 on isolation, loneliness and social connection, 2 on well-being, 2 on the use of digital tools, 2 on the fostering of socialization with peers.
  To evaluate the effects of the blended intervention and of the two conditions we will ask participants to fulfill the following clinical questionnaires: ULS-6 (Russell et al. 1980), MSPSS (Zimet et al., 1988), GAD-7 (Spitzer et al., 2006), PHQ-9 (Kroenke, Spitzer & Williams, 2001), SWLS (Diener et al., 1985), MLQ (Steger et al., 2006) before starting the intervention in presence and online (T0), at the end of that period (T1) and 2 months after (T2).
  Arms: intervention group

SUMMARY:
Extensive literature on social isolation and loneliness in young people points out that those conditions can negatively influence physical and psychological health, increasing the risks of loneliness-related health problems later in life. To date, especially after two years of the COVID-19 pandemic, the situation regarding loneliness and psychological frailties in young people has become even more urgent to address especially in populations at higher risks as for international students. This population in fact report to face greater social exclusion, discrimination, stigma, difficulties in cultural adaptation and more, compared to their peers, that can exacerbate loneliness and negatively impact on their psychological and physical health.

The pandemic delineated future directions for the development and implementation of digital interventions in the everyday clinical practice, many studies are starting to evaluate the efficacy and usability of blended (digital and in presence) psychological interventions within different populations. Thus, this study aims to assess the usability and efficacy of a blended psychosocial group intervention to tackle social isolation, loneliness and promoting well-being in this population.

DETAILED DESCRIPTION:
Rationale & background information:

Many studies have been conducted over the past two years regarding risks and challenges posed by the current situation towards youth frailties, psychological suffering, and social withdrawal derived from the pandemic. Some population are facing higher risks such as international college students that face difficulties such social isolation, loneliness and problems in getting in relationship with peers, with negative consequences on their wellbeing and mental health, as pointed out by different studies. Those difficulties have been enhanced by the pandemic as the social distancing, online classes and difficulties in adapting to a different context exacerbated many situations of vulnerability and resulted in severe clinical outcomes (anxiety, depression, mood disorders, loneliness health related outcomes, others).

Those scientific evidences underlined the importance of designing strategies of intervention to tackle those challenges fostering social inclusion, well-being empowerment and cultural adaptation in international students to prevent worse outcomes (such as immediate and long-term poor health outcomes, mental illnesses, increased suicidal risks) and to foster wellbeing and social connections.

Study goals:

The aim of this study is to investigate the impact and efficacy of a blended (in presence and online) psychosocial group intervention with peers in tackling social isolation, loneliness and empowering well-being in international college students.

Study design:

This study is a pilot randomized controlled trial of a blended (in presence and online) psychosocial group intervention.

Investigators anticipate recruiting a total of 30 participants that participated in the cross-sectional online survey and voluntarily left their email address to be recontacted to take part in the group activities. The participants will be randomly assigned into 2 groups with https://www.randomizer.org: experimental group (EG) composed of around 15 people and waiting list group (WG) composed of around 15 people. The participants of EG will take part in 8 psychosocial group sessions of 90 minutes each that will be held weekly between November 2022 and January 2023. The participants of WG will receive online self-help material regarding the same theme of the experimental group each week in the same period and will take part in the psychosocial group activities once the data collection will be over, approximately starting in March 2023. To evaluate the effects of the blended intervention and of the two conditions we will ask participants to fulfil clinical questionnaires (ULS-6, MSPSS, GAD-7, PHQ-9, SWLS, MLQ), before starting the intervention in presence and online (T0), at the end of that period (T1) and 2 months after (T2). The completion will take participants around 10 minutes.

Participants in the experimental group will fulfil the questionnaires pen-and-paper before the start of the group session, while participants in the control group will fulfil the questionnaires and the informed consent online through the use of qualtrics.com.

The psychosocial group intervention will consist of 8 sessions (one per week, duration estimated 90 minutes) that will be held in presence at the university clinical services. The themes that will be discussed during the sessions are related to social isolation, loneliness, well-being, mental health, tools to support connection with other peers and more.

Safety considerations:

The intervention will be conducted ensuring participants' physical and psychological safety, and no risks are identified during the intervention. To furtherly limit those risks, no potentially dangerous tools will be taken and used in the group activities (e.g. scissors, other dangerous objects).

Follow-up:

This study will include a follow-up with participants that will consist in the filling out of the clinical measures previously presented 2 months after the end of the intervention (experimental in presence intervention and online waiting list for the control group) to evaluate the long term effects of the intervention on well-being, loneliness and social support.

Data management:

All outcome measures of the experimental group will be recorded with pen-and-paper during the group session; on the contrary all outcome measures of the control group will be collected online through the use of qualtrics.com that will record their answers digitally. A research assistant will enter the data into an electronic database. A second research assistant independent from this study will check the quality and accuracy. The paper data collection sheets and signed informed consents will be stored in a locked cabinet, and the electronic database will be password-protected. The data will be kept confidential with only limited access to research investigators and related research assistants and graduate students.

Statistical analysis:

Investigators expect to use the paired-t test and analysis of covariance (ANCOVA) to analyze differences in baseline characteristics, baseline outcome measures and follow-up between the groups and determine the intervention effect for the 2 groups.

Qualitative analysis:

The study includes a qualitative evaluation of the personal experience and contents of the group activities proposed that will be collected through semi-structured interviews with participants at the end of the group intervention. A qualitative evaluation of the digital self-help materials provided online to both groups will be carried out with an online survey with close and open-ended questions to assess usability, accessibility and personal experience with the provided self-help materials and exercises.

Quality assurance:

The study was approved by the Ethics Committee of the School of Psychology at the University of Padua, protocol number 4800 (unique number: 06592A5FCBBFA818A5676B611295D2FC). The Committee will ensure that research is conducted according to the Declaration of Helsinki.

Problems anticipated:

The challenge for the study is the difficulty in recruiting participants. Recruiting international students facing social isolation and/or loneliness could be challenging. To address this problem, we will try to collaborate with other university services such as tutoring and mentoring services to inform their international student mentees about this study, as well as we will try to target international students who have enrolled to the university during the pandemic period and ask them to invite other international students they know via direct contact. This could lead to the inclusion (even if we will randomize participants) of some people that already know each other and or that already receive a form of support (social, practical etc.) that could empower and foster their well-being and socialization.

Project management:

The first and corresponding authors contribute to the study design, coordination, and project management. The first and second authors participate in the recruitment of participants, in the creation and delivery of the psychosocial intervention in presence and online. The first, second, and corresponding authors perform the data analyses, interpret them, draft and revise the manuscript. The corresponding author provided consultation throughout the entire process.

Ethics:

The study has approvals to send email invitations to participants based on data provided by students responding to a cross-sectional online survey and from other university services (e.g. tutoring and mentoring services).

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years,
* being an international student enrolled to a full university course at the University of Padua
* living in Padua
* Being able to communicate in English

Exclusion Criteria:

* Participants were excluded if they were Erasmus students
* not resident in Padua at the time of the intervention
* not responding to the invitation to participate in the group activities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Baseline before the group intervention (ULS-6) | the first week of intervention (T0)
  Participants of both groups (EG and CG) will fulfill the following measures to assess their baselines before the starting of the group intervention, objectives and clinical tools are the following:
  Loneliness will be assessed with ULS-6, short-form UCLA Loneliness Scale
Baseline before the group intervention (MSPSS) | the first week of intervention (T0)
  Participants of both groups (EG and CG) will fulfill the following measures to assess their baselines before the starting of the group intervention, objectives and clinical tools are the following:
  Perceived social support will be assessed with MSPSS, Multidimensional Scale of Perceived Social Support
Baseline before the group intervention (GAD-7) | the first week of intervention (T0)
  Participants of both groups (EG and CG) will fulfill the following measures to assess their baselines before the starting of the group intervention, objectives and clinical tools are the following:
  General Anxiety will be assessed with GAD-7, General Anxiety Disorder-7
Baseline before the group intervention (PHQ-9) | the first week of intervention (T0)
  Participants of both groups (EG and CG) will fulfill the following measures to assess their baselines before the starting of the group intervention, objectives and clinical tools are the following:
  General well-being will be assessed with PHQ-9, Patient Health Questionnaire-9
Baseline before the group intervention (SWLS) | the first week of intervention (T0)
  Participants of both groups (EG and CG) will fulfill the following measures to assess their baselines before the starting of the group intervention, objectives and clinical tools are the following:
  Psychological well-being will be assessed with SWLS, Satisfaction With Life Scale
Baseline before the group intervention (MLQ) | the first week of intervention (T0)
  Participants of both groups (EG and CG) will fulfill the following measures to assess their baselines before the starting of the group intervention, objectives and clinical tools are the following:
  Perception of personal well-being will be assessed with MLQ, Meaning in Life Questionnaire
Post intervention effect (from baseline to the last week of intervention) | the last week of the intervention (T1)
  Evaluation of change from the baseline (T0) to the last week of intervention (T1) in all the measures presented for (T0) baseline evaluation.
  Participants of both groups (EG and CG), at the end of the intervention (T1), will fulfill previously presented measures to assess changes from baseline (T0).
Follow up intervention effect (from baseline to follow up) | two months after the last week of the intervention (T2)
  Evaluation of change from the baseline (T0) to the follow up measurement 2 months after the end of the intervention (T2) in all the measures presented for (T0) baseline evaluation.
  Participants of both groups (EG and CG), at the follow up measurement 2 months after the end of the intervention (T2), will fulfill previously presented measures to assess changes from baseline (T0).
Follow up intervention effect (from last week of intervention to follow up) | two months after the last week of the intervention (T2)
  Evaluation of change from the post intervention (T1) to the follow up measurement 2 months after the end of the intervention (T2) in all the measures presented for (T0) baseline evaluation.
  Participants of both groups (EG and CG), at the follow up measurement 2 months after the end of the intervention (T2), will fulfill previously presented measures to assess changes from post intervention (T1).

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Cipolletta, PhD, Principal Investigator — University of Padova
Locations (1):
- SCUP - Servizi Clinici Universitari Psicologici, Padua, PD, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bu F, Steptoe A, Fancourt D. Who is lonely in lockdown? Cross-cohort analyses of predictors of loneliness before and during the COVID-19 pandemic. Public Health. 2020 Sep;186:31-34. doi: 10.1016/j.puhe.2020.06.036. Epub 2020 Aug 5. PMID 32768621
- [Background] Cipolletta S, Gris F. Older People's Lived Perspectives of Social Isolation during the First Wave of the COVID-19 Pandemic in Italy. Int J Environ Res Public Health. 2021 Nov 11;18(22):11832. doi: 10.3390/ijerph182211832. PMID 34831586
- [Background] Cipolletta, S., Mercurio, A., & Pezzetta, R. (2022). Perceived Social Support and Well-Being of International Students at an Italian University, Journal of International Students, 12(3). https://doi.org/10.32674/jis.v12i3.3954
- [Background] Cuijpers P, Auerbach RP, Benjet C, Bruffaerts R, Ebert D, Karyotaki E, Kessler RC. The World Health Organization World Mental Health International College Student initiative: An overview. Int J Methods Psychiatr Res. 2019 Jun;28(2):e1761. doi: 10.1002/mpr.1761. Epub 2019 Jan 6. PMID 30614123
- [Background] Haikalis M, Doucette H, Meisel MK, Birch K, Barnett NP. Changes in College Student Anxiety and Depression From Pre- to During-COVID-19: Perceived Stress, Academic Challenges, Loneliness, and Positive Perceptions. Emerg Adulthood. 2022 Apr;10(2):534-545. doi: 10.1177/21676968211058516. PMID 35382515
- [Background] Karyotaki E, Cuijpers P, Albor Y, Alonso J, Auerbach RP, Bantjes J, Bruffaerts R, Ebert DD, Hasking P, Kiekens G, Lee S, McLafferty M, Mak A, Mortier P, Sampson NA, Stein DJ, Vilagut G, Kessler RC. Sources of Stress and Their Associations With Mental Disorders Among College Students: Results of the World Health Organization World Mental Health Surveys International College Student Initiative. Front Psychol. 2020 Jul 30;11:1759. doi: 10.3389/fpsyg.2020.01759. eCollection 2020. PMID 32849042
- [Background] Song B, Zhao Y, Zhu J. COVID-19-related Traumatic Effects and Psychological Reactions among International Students. J Epidemiol Glob Health. 2021 Mar;11(1):117-123. doi: 10.2991/jegh.k.201016.001. Epub 2020 Oct 24. PMID 33605116